CLINICAL TRIAL: NCT02553551
Title: Effect of Vitamin C on Postoperative Pain After Laparoscopic Cholecystectomy; a A Prospective Randomized Controlled Trial
Brief Title: Effect of Vitamin C on Postoperative Pain After Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taeho Hong (Other)
Responsible Party: Sponsor-Investigator, Taeho Hong, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Seoul-06
Record Dates: First submitted 2015-09-13; First posted 2015-09-17 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Cholecystitis; Cholelithiasis
MeSH Terms: conditions — Cholelithiasis | interventions — Ascorbic Acid; Vitamins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin C (Experimental): During the period of hospitalization, Intake of vitamin C 3000 mg per day via oral route until the day of discharge.
  After discharge, no additional vitamin C pill was given.
  Interventions: Drug: Vitamin C
- Placebo (Placebo Comparator): During the period of hospitalization, Intake of gelatinous capsule three times per day via oral route until the day of discharge.
  After discharge, no additional capsule was given.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin C — During the period of hospitalization, Intake of vitamin C 3000 mg per day via oral route until the day of discharge.
  After discharge, no additional vitamin C pill was given.
  Other Names: Vitamin
  Arms: Vitamin C
Drug: Placebo — During the period of hospitalization, Intake of gelatinous capsule three times per day via oral route until the day of discharge.
  After discharge, no additional capsule was given.
  Other Names: placebo capsule
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the effect of Vitamine C supplements to be helpful to reduce the postoperative pain after laparoscopic cholecystectomy through the double-blinded randomized controlled trial.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of Vitamine C supplements to be helpful to reduce the postoperative pain after laparoscopic cholecystectomy through the double-blinded randomized controlled trial.

The primary purpose of this study is to confirm the reduce of postoperative pain through the oral supplement of Vitamine C before and after the surgery. For this purpose, we compared the dosage or counts of opioids usage with the oral supplement of Vitamine C or not.

The secondary purpose is to assess the pain score, postoperative morbidities, postoperative length of stay or postoperative time between two groups.

ELIGIBILITY:
Inclusion Criteria:

* chronic cholecystitis
* gallbladder polyp

Exclusion Criteria:

* grade I Tokyo guideline for acute cholecystitis
* grade II Tokyo guideline for acute cholecystitis without the evidence of gallbladder perforation
* gallbladder cancer
* the patient who underwent reduced port surgery
* the patient who underwent common bile duct exploration during the operation
* the patient who underwent concurrent operation
* the patient who had past history of upper abdominal surgery
* the patient who had a immunodeficiency state
* the case which had a suspicion of delayed bile leakage
* the case which had a incomplete cystic duct ligation
* the patient who underwent open conversion surgery during the operation
* the patient who had a high risk of bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The postoperative pain | The change of pain score between 6hours after operation and 24hours after operation
  Postoperative pain was estimated using the visual analog scale (VAS) from 0 (no pain) to 10 (worst pain imaginable) at 6, 24, and 48 hours after the operation.

SECONDARY OUTCOMES:
Postoperative morbidity | 30 days
  the incidence of complications after surgery during one month after surgery such as postoperative fever, atelectasis, infectious complications, bile leak, postoperative bleeding, readmission or mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Taeho Hong, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Department of HBP Surgery, Seoul St. Mary's hospital, Seoul, Seocho-gu, Banopo-dong, South Korea